CLINICAL TRIAL: NCT06304454
Title: Board Games at Kindergarten (5 Years Old) to Improve Cognitive and Emotional Processes
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brain In Game scientific-technical service (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: P5_BG
Record Dates: First submitted 2024-02-29; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Kindergarten Children
Keywords: Cognitive change; Emotional change; Child development; Kindergarten

STUDY DESIGN:
Intervention Model Description: Cluster RCT
Who Masked: Participant, Outcomes Assessor
Masking Description: Double (outcomes assessor and participants)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive and emotional board games (Experimental): An experimental group that will carry out the cognitive and emotional game program in the classroom implemented by the teachers of the participating centers.
  Interventions: Other: Board game intervention
- Motor/Luck board games (Active Comparator): A control group that will be on board games that do not directly activate cognitive and emotional processes. These games are classified as motor or luck board games.
  Interventions: Other: Board game intervention

INTERVENTIONS:
Other: Board game intervention — 5 weeks / 2 sessions each week / 1 hour each session

SUMMARY:
Cognitive (i.e. executive functions, memory) and socio-emotional (i.e. affection recognition) processes emerges at first years. These processes have been frequently related to adequate academic performance in the scientific literature (Passolunghi et al, 2015). Current research aimed at training cognitive processes found promising results using board game as a cognitive tool in children (Passolunghi & Costa, 2016). Considering the growing interest of teachers in this playful and possibly educational, cognitive and socio-emotional resource, a game program for these purposes has been designed to be used in kindergarten classrooms.

The main aim of the present study is to test the efficacy of a cognitive and emotional training program in the classroom based on board games in kindergarten students (5 years old). For this, there will be an experimental group that will carry out the cognitive and emotional game program in the classroom implemented by the teachers of the participating centers, and a control group that will be on board games that do not directly activate cognitive and emotional processes. At the end of the interventions, the groups will be compensated by carrying out inversely both board game programs. The classes will be randomly assigned to an experimental group and a passive control group.

DETAILED DESCRIPTION:
The hypothesis from this study are: i) the experimental group will show a significantly greater improvement in the neuropsychological tasks that measure cognitive and emotional processes compared to the active control group after the intervention; ii) the experimental group will show a significantly greater improvement in the tests evaluated by their parents after the intervention compared to the active control group. All hypotheses will be controlled for age and socioeconomic status.

ELIGIBILITY:
Inclusion Criteria:

* To be enrolled in an ordinary educational center.
* To provide informed consent from both parents and the participant's agreement to participate in the study.

Exclusion Criteria:

• Sensory/comprehension difficulties that make it impossible to carry out the program activities.

Ages: 5 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-03-15 (Estimated)

PRIMARY OUTCOMES:
Visual Memory | Baseline and Post-intervention (after 5 weeks)
  Change in visual memory from baseline to post intervention. The task to assess visual memory is the subtest Picture Memory from the WPPSI-IV. This subtest consists of the child viewing a stimulus page of pictures for a specified time and then to select those same pictures from the options given. When the response is correct was scored 1, and 0 when incorrect. The task finished when the child made 3 consecutive mistakes. The total score is the sum of scores on Items 1-35, which ranged from 0 to 35.
Processing speed and inhibition | Baseline and Post-intervention (after 5 weeks)
  Change in processing speed and inhibition from baseline to post intervention. The task used to assess these outcomes is included in the neuropsychological battery NEPSY-II. The task Naming and Inhibition consists of two blocks: a series of white and black shapes (circles and squares) and a series of arrows with different directions (up and down). The first part of each block is the task of shape/direction naming (in this case, a child had to name the shapes/direction he/she saw) at a rapid pace and the inhibition task. The second part if the inhibition task, in which the child need to change the rule: if he/she saw a square, he/she was to say "circle " and so forth or if he/she saw an up direction, need to say down. Each task record the number of corrected/non-corrected mistakes and the amount of time the child spent doing each task.
Affect recognition | Baseline and Post-intervention (after 5 weeks)
  Change in affect recognition from baseline to post intervention. This subtest from the NEPSY-II assesses a child's ability to recognize six different emotional expressions (happiness, sadness, anger, disgust, fear, and a neutral expression) from photographs of children's faces in different tasks (select two photographs with identical affect from 3 or 4; select one of the four photographs that depicted identical affect as a photograph at the top of a page in the stimulus book). When the response is correct was scored 1, and 0 when incorrect. The total score is the sum of scores on Items 1-25, which ranged from 0 to 25. This subtest also gave the total of incorrect responses for each emotion.

SECONDARY OUTCOMES:
Hollingshead Index (Hollingshead, 1975) | Baseline
  Sociodemographic data (age, sex, school year and socioeconomic status)
CHEXI (Giménez et al. 2022) | Baseline and Post-intervention (after 5 weeks)
  Change in common behavioral executive functions from baseline to post intervention.
  The test consists of 24 items with 5 response options ranging from 1 (Definitely not true) to 5 (Definitely true). Two factors have been considered: WM and Inhibition. In this study, responders are the parents of the children. Higher ratings mean poor executive functioning.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Education, Psychology and Social Work; University of Lleida, Lleida, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Passolunghi MC, Costa HM. Working memory and early numeracy training in preschool children. Child Neuropsychol. 2016;22(1):81-98. doi: 10.1080/09297049.2014.971726. Epub 2014 Nov 4. PMID 25366543
- [Background] Passolunghi MC, Lanfranchi S, Altoe G, Sollazzo N. Early numerical abilities and cognitive skills in kindergarten children. J Exp Child Psychol. 2015 Jul;135:25-42. doi: 10.1016/j.jecp.2015.02.001. Epub 2015 Mar 25. PMID 25818537
- [Background] Giménez, A., López-Zamora, M., Vila, O., Sánchez, A., & Thorell, L. B. (2022). Fiabilidad y validez de la versión española del
- [Background] Hollingshead, A. B. (1975). Four factor index of social status. Retrieved from: https://sociology.yale.edu/sites/default/files/files/yjs_fall_2011.pdf#page=21
- [Background] Korkman, M., Kirk, U., & Kemp, S. (2007). NEPSY-II (2nd Ed.). San Antonio: Pearson PsychCorp.
- [Background] Wechsler, D. (2014). WPPSI-IV, Escala de Inteligencia de Wechsler para preescolar y primaria (4th Ed.). Madrid/Barcelona: Pearson Clinical Assessment Spain.